CLINICAL TRIAL: NCT02379858
Title: Gastrointestinal Tract Recovery in Patients Undergoing Open Ventral Hernia Repair: A Multi-Center, Randomized, Double-Blind, Trial of Alvimopan and Placebo
Brief Title: Gastrointestinal Tract Recovery in Patients Undergoing Open Ventral Hernia Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer of Alvimopam closed the study due to low enrollment.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Matthew I. Goldblatt, Director, Condon Hernia Institute, Associate Professor of Surgery, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO24196
Record Dates: First submitted 2015-02-21; First posted 2015-03-05 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Ventral Hernia
Keywords: GI Tract Recovery; Hospital Discharge
MeSH Terms: conditions — Hernia, Ventral | interventions — alvimopan; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alvimopan (Entereg) (Experimental): Alvimopan, 12mg, capsule. One 30 to 90 minutes before the scheduled start of surgery on Day 0, and twice daily beginning on POD 1 after NGT removal until hospital discharge or for a maximum of 7 days (up to 15 doses) of postoperative treatment. First post-operative dose begins after NGT removal.
  Interventions: Drug: Alvimopan
- Suger Pill (Control) (Placebo Comparator): Placebo, 12mg capsule. One 30 to 90 minutes before the scheduled start of surgery on Day 0, and twice daily beginning on POD 1 until hospital discharge or for a maximum of 7 days (up to 15 doses) of postoperative treatment. First post-operative dose begins after NGT removal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan — Alvimopan, 12mg, capsule. One 30 to 90 minutes before the scheduled start of surgery on Day 0, and twice daily beginning on POD 1 after NGT removal until hospital discharge or for a maximum of 7 days (up to 15 doses) of postoperative treatment. First post-operative dose begins after NGT removal.
  Other Names: Entereg
  Arms: Alvimopan (Entereg)
Drug: Placebo — Placebo (sugar pill-will be the same size and color as the Alvimopan capsule), 12mg capsule. One 30 to 90 minutes before the scheduled start of surgery on Day 0, and twice daily beginning on POD 1 until hospital discharge or for a maximum of 7 days (up to 15 doses) of postoperative treatment. First post-operative dose begins after NGT removal.
  Other Names: Sugar Pill
  Arms: Suger Pill (Control)

SUMMARY:
The purpose of this study is to determine whether Alvimopan (Entereg) in ventral hernia surgery patients is associated with accelerated gastrointestinal recovery and reduced length of hospital stay compared to placebo controls.

DETAILED DESCRIPTION:
Background: One of the most common occurrences following ventral incisional hernia repair is post-operative ileus. Post-operative ileus is a source of patient discomfort and morbidity that ultimately delays discharge from the hospital and is frequently a source of patient readmission. Prolonged length of hospital stay due to post-operative ileus increases direct health care costs, as well as the indirect costs of a delay in returning to the workforce. The cause of prolonged ileus is multifactorial, but some of the main culprits include intra-operative bowel manipulation, the release of endogenous opioids, the administration of exogenous opioid analgesics during surgery and for post-operative pain control, inflammation, and fluid shifts. A study by Lowe et al showed that following ventral hernia repair, 27% of their study patients had a prolonged ileus, defined as lasting more than 7 days postoperatively. Likewise, the mean hospital stay for these patients was 12.5 days, due most frequently, to a delayed return of bowel function.

Ventral incisional hernia repair is a common operation and post-operative ileus remains a frequent and costly post-operative occurrence for which we do not currently have an effective therapy. Alvimopan has proven to successfully decrease the duration of post-operative ileus and is FDA approved for such use in patients who have undergone bowel resection. Ultimately, decreasing the interlude between operation and return of bowel function results in shorter hospital stays, lower hospital costs, and faster rehabilitation. We propose to study the effectiveness of Alvimopan in decreasing postoperative ileus time in patients undergoing ventral hernia repair, a cohort that we feel may benefit from the use of Alvimopan but that to date has not been studied.

Recruitment and Sample Size: A total of 140 patients are expected to undergo research related treatments. The study will contain one open surgery arm. The open surgery arm will be a single-site prospective, randomized, double-blinded, placebo-controlled clinical trial with 1:1 randomization between the study drug and placebo with 70 patients in each group for a total of 140 patients in the study. An interim evaluation of efficacy will be conducted separately in the open surgery arm when half the patients have been recruited.

This study is expected to enroll up to 140 subjects from one academic medical center (Froedtert Hospital and the Medical College of Wisconsin) a site that performs state of the art hernia repairs and is a high volume hernia practices.

Treatment: Consented patients in the Treatment Group will receive 12 milligrams (mg) of Alvimopan per-oral (PO) 30 to 90 minutes prior to ventral hernia repair in the pre-operative area and continue 12 mg PO twice daily until hospital discharge or post-operative day (POD) 7 for a maximum of 15 in-hospital doses (Appendix II). The first post-operative dose will begin after Nasogastric Tube (NGT) removal.

Patients in the Control Group will receive 12 milligrams (mg) of Placebo orally (PO) 30 to 90 minutes prior to Ventral Hernia Repair (VHR) in the pre-operative area and continue 12 mg PO twice a day until hospital discharge or post-operative (POD) 7 for a maximum of 15 in-hospital doses. The first post-operative dose will begin after NGT removal.

Warnings and precautions as provided in the prescribing information packet and US PI include:

1. A higher number of myocardial infarctions was reported in patients treated with alvimopan 0.5 mg twice daily compared with placebo 12 in a 12-month study in patients treated with opioids for chronic pain, although a causal relationship has not been established
2. Patients recently exposed to opioids are expected to be more sensitive to the effects of ENTEREG and therefore may experience abdominal pain, nausea and vomiting, and diarrhea.
3. Not recommended in patients with severe hepatic impairment.
4. Not recommended in patients with end stage renal disease.
5. Most common adverse reaction (incidence >=1.5%) occurring with a higher frequency than placebo among ENTEREG-treated patients undergoing surgeries that included a bowel resection was dyspepsia [2013 PI].
6. Not recommended in patients with complete GI obstruction or in patients who have surgery for correction of complete bowel obstruction.
7. Not recommended in pancreatic or gastric anastomosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be informed about the study, have read, understood, and signed the Informed Consent Form
2. Subjects of either gender that are ≥18 years of age
3. Subjects who can ambulate preoperatively
4. Subjects will have a Body-Mass Index (BMI) of ≤ 40mg/m2
5. Subjects with an American Society of Anesthesiologists (ASA) classification of 1, 2 or 3
6. Subjects not receiving an epidural to control perioperative pain
7. Subjects will be undergoing elective single-staged open ventral (incisional or midline) hernia repair
8. Subjects in which intra-operatively their surgical field/wound is characterized as Type 1 (Appendix II)
9. Subjects with a hernia defect ≥9 cm2 large

Exclusion Criteria:

1. Subjects who are not able to comprehend or comply with study requirements
2. Subjects who are pregnant
3. Subjects with BMI > 40
4. Subjects with autoimmune disorder requiring >10mg of a corticosteroid per day
5. Subjects with pre-existing systemic infections
6. Subjects with a wound-healing disorder
7. Subjects who have taken therapeutic doses of opioids for more than 7 consecutive days immediately prior to taking Alvimopan
8. Subjects who are immunocompromised such as HIV or transplant, or receiving chemo or radiation therapy
9. Subjects with a hernia defect < 9cm2 large when measured intra-operatively
10. Subjects in which intra-operatively their surgical wound field/wound is characterized as Type 2, 3, or 4 (Appendix II)
11. Subjects in which the ventral incisional hernia repair requires more than one operation to reduce the hernia or to complete the hernia repair
12. Subjects with a hernia repair requiring an emergent procedure
13. Subjects in which untreated cancer was found intra-operatively
14. Subjects with cirrhosis or are currently being treated with dialysis
15. Subjects with severe hepatic impairment (Childs-Pugh class C)
16. Subjects with end-stage renal disease
17. Subjects scheduled for a concomitant procedure that involves the GI tract
18. Subjects with unplanned procedures that involve the GI tract
19. Subjects requiring post-operative NGT
20. Subjects participating in another prospective interventional study that involves the use of a device, drug, or surgery that would compromise the current study
21. Subjects with an epidural to control perioperative pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew I Goldblatt, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger D, Bientzle M, Muller A. Postoperative complications after laparoscopic incisional hernia repair. Incidence and treatment. Surg Endosc. 2002 Dec;16(12):1720-3. doi: 10.1007/s00464-002-9036-y. Epub 2002 Sep 6. PMID 12209325
- [Background] Buchler MW, Seiler CM, Monson JR, Flamant Y, Thompson-Fawcett MW, Byrne MM, Mortensen ER, Altman JF, Williamson R. Clinical trial: alvimopan for the management of post-operative ileus after abdominal surgery: results of an international randomized, double-blind, multicentre, placebo-controlled clinical study. Aliment Pharmacol Ther. 2008 Aug 1;28(3):312-25. doi: 10.1111/j.1365-2036.2008.03696.x. PMID 19086236
- [Background] Delaney CP, Wolff BG, Viscusi ER, Senagore AJ, Fort JG, Du W, Techner L, Wallin B. Alvimopan, for postoperative ileus following bowel resection: a pooled analysis of phase III studies. Ann Surg. 2007 Mar;245(3):355-63. doi: 10.1097/01.sla.0000232538.72458.93. PMID 17435541
- [Background] Lowe JB 3rd, Lowe JB, Baty JD, Garza JR. Risks associated with "components separation" for closure of complex abdominal wall defects. Plast Reconstr Surg. 2003 Mar;111(3):1276-83; quiz 1284-5; discussion 1286-8. doi: 10.1097/01.PRS.0000047021.36879.FD. PMID 12621202
- [Background] Ludwig K, Enker WE, Delaney CP, Wolff BG, Du W, Fort JG, Cherubini M, Cucinotta J, Techner L. Gastrointestinal tract recovery in patients undergoing bowel resection: results of a randomized trial of alvimopan and placebo with a standardized accelerated postoperative care pathway. Arch Surg. 2008 Nov;143(11):1098-105. doi: 10.1001/archsurg.143.11.1098. PMID 19015469
- [Background] McGreevy JM, Goodney PP, Birkmeyer CM, Finlayson SR, Laycock WS, Birkmeyer JD. A prospective study comparing the complication rates between laparoscopic and open ventral hernia repairs. Surg Endosc. 2003 Nov;17(11):1778-80. doi: 10.1007/s00464-002-8851-5. Epub 2003 Sep 10. PMID 12958679
- [Background] Vargo D. Component separation in the management of the difficult abdominal wall. Am J Surg. 2004 Dec;188(6):633-7. doi: 10.1016/j.amjsurg.2004.08.051. PMID 15619476
- [Background] Wolff BG, Michelassi F, Gerkin TM, Techner L, Gabriel K, Du W, Wallin BA; Alvimopan Postoperative Ileus Study Group. Alvimopan, a novel, peripherally acting mu opioid antagonist: results of a multicenter, randomized, double-blind, placebo-controlled, phase III trial of major abdominal surgery and postoperative ileus. Ann Surg. 2004 Oct;240(4):728-34; discussion 734-5. doi: 10.1097/01.sla.0000141158.27977.66. PMID 15383800
- [Background] Wolff BG, Weese JL, Ludwig KA, Delaney CP, Stamos MJ, Michelassi F, Du W, Techner L. Postoperative ileus-related morbidity profile in patients treated with alvimopan after bowel resection. J Am Coll Surg. 2007 Apr;204(4):609-16. doi: 10.1016/j.jamcollsurg.2007.01.041. PMID 17382220
- [Background] Itawi EA, Savoie LM, Hanna AJ, Apostolides GY. Alvimopan addition to a standard perioperative recovery pathway. JSLS. 2011 Oct-Dec;15(4):492-8. doi: 10.4293/108680811X13176785204076. PMID 22643504
- [Background] Poulose BK, Shelton J, Phillips S, Moore D, Nealon W, Penson D, Beck W, Holzman MD. Epidemiology and cost of ventral hernia repair: making the case for hernia research. Hernia. 2012 Apr;16(2):179-83. doi: 10.1007/s10029-011-0879-9. Epub 2011 Sep 9. PMID 21904861

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alvimopan (Entereg) | Suger Pill (Control)
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan (Entereg) | Suger Pill (Control) | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.7) | 69.2 (3.8) | 60 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Length of Time (Hrs/Days) to Gastrointestinal Tract Recovery
Description: Time to gastrointestinal recovery will be measured by the following:
  Time to first flatus and time to first bowel movement measured twice daily. Toleration of a diet and toleration of oral pain medication defined as ingestion of diet or medications that occurs without vomiting or significant nausea for four hours following ingestion.
  GI-2 recovery defined as both toleration of solid food and occurrence of first bowel movement. GI-3 recovery is defined as toleration of solid food and either occurrence of first flatus or occurrence of first bowel movement.
  Patients requiring nasogastric tube insertion, requiring reduction or restriction of diet, having episodes of emesis, and/or needing initiation of Total Parenteral Nutrition (TPN) will be recorded. VAS (visual analog pain scale), nausea, and bloating will be recorded by nursing staff at least twice daily. The number of doses of anti-nausea medication administered during the hospitalization will also be recorded.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 week.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Alvimopan (Entereg) | Suger Pill (Control)
Number analyzed (Participants) | 6 | 4
Days | 2.8 (1.3) | 3.5 (1)

2. Secondary Outcome: Length of Hospital Stay
Description: Length of stay will be measured in hours from the time that surgery is completed until the hospital discharge order is written (hrs/days).
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Alvimopan (Entereg) | Suger Pill (Control)
Number analyzed (Participants) | 6 | 4
Days | 4.7 (1.5) | 5 (1.4)

3. Secondary Outcome: 30-day Treatment Related Morbidity and Re-admission Rates
Description: Treatment (study drug) and surgery (complications as a direct result of surgery) related morbidity and re-admission rates will be assessed from the time surgery is completed to 30-days post-operatively. Treatment related morbidity and re-admission rates include: post-operative ileus (POI), indigestion and any event determined by the attending physician to be directly related to treatment (study drug). Surgical complications include: hernia recurrence, infections, and any event determined by the attending physician to be directly related to surgery.
Time Frame: Participants will be followed for the duration of hospital stay to 30 days after surgery, an expected average of 6 weeks
Measure: Mean (Standard Deviation); unit: morbidity or readmission
Arm/Group | Alvimopan (Entereg) | Suger Pill (Control)
Number analyzed (Participants) | 6 | 4
morbidity or readmission | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Followed clinicaltrials.gov definitions.
Arm/Group | Alvimopan (Entereg) | Suger Pill (Control)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT02379858/Prot_SAP_000.pdf